CLINICAL TRIAL: NCT02890082
Title: Pilot Study of Preservation of Fertility by Ovarian Stimulation Associated With Tamoxifen, and Freezing Oocyte or Embryo Prior Chemotherapy for Breast Cancer
Brief Title: Preservation of Fertility by Ovarian Stimulation Associated With Tamoxifen, Prior Chemotherapy for Breast Cancer
Acronym: PRESAGE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICO-N-2013-03
Record Dates: First submitted 2016-08-26; First posted 2016-09-07 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; fertility; chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Luteal Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tamoxifen stim in early follicular phase (Experimental): Day cycle of the patient when ovarian stimulation begin (early follicular phase) = D1 to D3
  Interventions: Drug: Tamoxifen stim in early follicular phase
- Tamoxifen stim in late follicular phase (Other): Day cycle of the patient when ovarian stimulation begin (late follicular phase) = D4 to D14
  Interventions: Drug: Tamoxifen stim in late follicular phase
- Tamoxifen stim in luteal phase (Other): Day cycle of the patient when ovarian stimulation begin (luteal phase) = D15 to D28
  Interventions: Drug: Tamoxifen stim in luteal phase

INTERVENTIONS:
Drug: Tamoxifen stim in early follicular phase — Day cycle of the patient when ovarian stimulation begin (early follicular phase) = D1 to D3
  * Stimulation with simultaneously: TAM (tamoxifen) 60mg / day + FSH® 150 to 300 IU / day (following ovarian reserve)
  * Monitoring (ultrasound + blood test E2, LH (luteinizing hormone) and P) every 2 to 3 days +/- dose adjustment of FSH
  * Ovulation by blocking the GnRH antagonist (gonadotropin-releasing hormone : CETROTIDE) introduced according to the usual criteria,
  * Continued monitoring (ultrasound + blood test E2, LH and P) every 2 to 3 days
  * Triggering ovulation by OVITRELLE ® 250μg according to the usual criteria
  * 35 h after the onset, oocyte puncture transvaginally the gynecology unit under local or general anesthesia.
  Other Names: Hormotherapy
  Arms: Tamoxifen stim in early follicular phase
Drug: Tamoxifen stim in late follicular phase — Day cycle of the patient when ovarian stimulation begin (late follicular phase) = D4 to D14
  * Monitoring (ultrasound + blood test E2, LH and P) until a follicle of 15 mm
  * Ovulation induction by OVITRELLE® 250μg.
  * Continued monitoring (ultrasound + blood test E2, LH and P) 4 days after OVITRELLE® to the proper stage for the beginning of stimulation.
  * Stimulation with simultaneously: TAM 60mg / day + FSH® 150 to 300 IU / day (following ovarian reserve) + CETROTIDE
  * Continued monitoring (ultrasound + blood test E2, LH and P) every 2 to 3 days +/- adaptation of FSH
  * Triggering ovulation by OVITRELLE ® 250μg according to the usual criteria
  * 35 h after the onset, oocyte puncture transvaginally the gynecology unit under local or general anesthesia.
  Other Names: Hormotherapy
  Arms: Tamoxifen stim in late follicular phase
Drug: Tamoxifen stim in luteal phase — Day cycle of the patient when ovarian stimulation begin (luteal phase) = D15 to D28
  * 1 or 2 Monitoring (ultrasound + blood test E2, LH and P) to check the validity of the post-ovulatory phase
  * Stimulation with simultaneously: TAM 60mg / day + FSH® 150 to 300 IU / day (following ovarian reserve) + CETROTIDE
  * Continued monitoring (ultrasound + blood test E2, LH and P) every 2 to 3 days +/- adaptation of FSH
  * Triggering ovulation by OVITRELLE ® 250μg according to the usual criteria
  * 35 h after the onset, oocyte puncture transvaginally the gynecology unit under local or general anesthesia
  Other Names: Hormotherapy
  Arms: Tamoxifen stim in luteal phase

SUMMARY:
The rates of patients with spontaneous pregnancies reported after breast cancer is between 3 and 7%, particularly because of these treatments.

Therefore, it is essential to anticipate this problem by proposing the use of fertility preservation techniques for these young patients prior to any gonadotoxic treatment.

PRESAGE study offers to patients fewer than 40, to preserve their fertility before neoadjuvant or adjuvant chemotherapy for invasive breast cancer.

The aim of this study is to evaluate the feasibility of ovarian stimulation emergency order not to delay the start of treatment. This stimulation combined gonadotropin and tamoxifen followed by an oocyte retrieval. The patient may receive an oocyte vitrification and / or embryonic.

This procedure is already done in many countries, and by some French teams, by combining tamoxifen or letrozole to the classic gonadotropin stimulation.

DETAILED DESCRIPTION:
With 50 000 new cases per year, breast cancer is the most common cancer in women in France. About a quarter of breast cancers occurs before menopause and 7% before the age of 40 years. Due to the increased incidence of breast cancer in young women and declining age of first pregnancy, it is not unusual to have patient desiring pregnancy after treatment of a breast cancer. Among these women, the use of adjuvant therapy (chemotherapy, hormone therapy, chemical castration) is common. Adjuvant or neoadjuvant chemotherapy resulted in significantly lower recurrence rates and increase the survival of these patients, but these treatments could have more or less long-term consequences, including in ovarian function. Ovarian consequences of these therapeutic must also be explained to young patients. But it seems that this information is often inadequate or poorly understood, and then patients deplore to be faced with secondary infertility.

The rates of patients with spontaneous pregnancies reported after breast cancer is between 3 and 7%, particularly because of these treatments.

Therefore, it is essential to anticipate this problem by proposing the use of fertility preservation techniques for these young patients prior to any gonadotoxic treatment.

PRESAGE study offers to patients fewer than 40, to preserve their fertility before neoadjuvant or adjuvant chemotherapy for invasive breast cancer.

The aim of this study is to evaluate the feasibility of ovarian stimulation emergency order not to delay the start of treatment. This stimulation combined gonadotropin and tamoxifen followed by an oocyte retrieval. The patient may receive an oocyte vitrification and / or embryonic.

This procedure is already done in many countries, and by some French teams, by combining tamoxifen or letrozole to the classic gonadotropin stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40
* infiltrating breast carcinoma histologically proven
* Indication of adjuvant or neoadjuvant chemotherapy
* T0-T1-T2-T3
* N0-N1-N2a
* M0 after staging
* AMH ≥1 ng / mL and / or account antral follicles ≥ 5
* HIV serology negative.

Exclusion Criteria:

* breast cancer history
* History of another cancer in the last 5 years, with the exception of basal cell skin cancer and squamous cell
* patient in pregnancy
* pulmonary embolism under 6 months
* deep vein thrombosis of less than 6 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of ovarian stimulation combining tamoxifen with recombinant FSH (follicle stimulating hormone ) followed by oocyte vitrification and / or embryo freezing before chemotherapy for breast cancer. | max 1 month after beginning of stimulation (At the end of oocyte puncture after ovarian stimulation)
  Assess the feasibility of ovarian stimulation combining tamoxifen with recombinant FSH (follicle stimulating hormone ) followed by oocyte vitrification and / or embryo freezing before chemotherapy for breast cancer.
  => evaluated by number of oocytes and / or embryos per patient.

SECONDARY OUTCOMES:
number of pregnancy obtain | At least 2 years After chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: BORDES Virginie, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- ICO René Gauducheau, Nantes, France

IPD SHARING:
Plan to Share IPD: No